CLINICAL TRIAL: NCT01103037
Title: A Randomized, Double-blind, Parallel Group Study to Compare the Pharmacodynamics/Efficacy, Safety and Pharmacokinetics of QAV680 Versus Placebo in Patients With Moderate Persistent Asthma
Brief Title: Efficacy, Safety and Pharmacokinetics of QAV680 Versus Placebo in Patients With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAV680A2201E1; 2009-017267-41 (EudraCT Number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Asthma
Keywords: Mild; Moderate; Asthma
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — NVP-QAV680

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- QAV680 (Experimental)
  Interventions: Drug: QAV680
- QAV680 Placebo (Placebo Comparator)
  Interventions: Drug: QAV680 Placebo

INTERVENTIONS:
Drug: QAV680 — QAV680 500 mg (5 x 100 mg capsules) four times per day
  Arms: QAV680
Drug: QAV680 Placebo — Placebo to QAV680 5 capsules four times per day
  Arms: QAV680 Placebo

SUMMARY:
This study will assess the safety and efficacy of QAV680 in patients with mild to moderate asthma

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate persistent asthma

Exclusion Criteria:

* Smokers
* Any significant disease or illness, other than asthma

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in one second (FEV1) as measured by Spirometry | 28 days

SECONDARY OUTCOMES:
FEV1 assessments at various timepoints including time of peak drug concentration | 28 days
Measure the change in exhaled Nitric Oxide (FeNO) | 28 days
Assessment of the pharmacokinetics of multiple doses of QAV680 in patients with mild to moderate asthma. | 28 days
Total serum IgE levels | 28 days
Change in daily variability in the morning and evening Peak Expiratory Flow Rate (PEFR) from Baseline. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (3):
  - West Coast Clinical Trials, Cypress, California
  - American Health Research, Charlotte, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Results for CQAV680A2201E1 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6683